CLINICAL TRIAL: NCT03649308
Title: Negative Pressure Wound Therapy Compared to Traditional Care After Split-thickness Skin Grafting - a Randomized Controlled Trial
Brief Title: Negative Pressure Wound Therapy Compared to Traditional Care After Skin Grafting
Acronym: TRUTH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Finland Hospital District (Other)
Collaborators: Tampere University Hospital (Other); University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6U/2018
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Wound of Skin; Wound Heal; Wound; Wound Open; Wound Breakdown; Skin Wound; Skin Scarring
Keywords: Negative pressure wound therapy; Skin graft; split-thickness skin graft
MeSH Terms: conditions — Wounds and Injuries; Surgical Wound Dehiscence; Cicatrix | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: After split-thickness skin graft procedure, the participants are assigned to either conventional treatment or negative pressure wound therapy group in parallel for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Negative Pressure Wound Therapy (Experimental): A negative pressure wound therapy device (PICO) is applied on split-thickness skin graft for 5 to 7 days from surgery in operating theatre. The patient can be mobilized immediately after skin graft procedure.
  Interventions: Device: Negative Pressure Wound Therapy
- Conventional treatment (Active Comparator): A conventional wound dressing is applied on wound in operating theatre, followed by immobilization for 5 days after split-thickness skin graft procedure.
  Interventions: Procedure: Conventional treatment

INTERVENTIONS:
Device: Negative Pressure Wound Therapy — An immediate mobilization and negative pressure wound therapy (PICO) initiated after surgery.
  Arms: Negative Pressure Wound Therapy
Procedure: Conventional treatment — Traditional treatment with conventional wound dressing and 5 days of immobilization after surgery.
  Arms: Conventional treatment

SUMMARY:
The aim of this study is to compare negative pressure wound therapy to traditional care after split-thickness skin grafting in patients aged over 18.

DETAILED DESCRIPTION:
Split-thickness skin grafting (STSG) is one of the most commonly used techniques in reconstructive plastic surgery and dermatology. Skin grafts are being used to cover skin defects caused by multiple etiologies. Traditionally, patients are immobilized in bed or in wheelchair for up to five days after surgery. Long immobilization decreases patients overall ability to function and increases the length of the stay in hospital. Negative pressure wound therapy (NPWT) have been used successfully in treatment of acute, chronic and diabetic ulcers. It is proposed that NPWT increases capillary blood flow, decreases bacterial contamination, seroma formation and swelling. Using NPWT on split-thickness skin grafts after burns is well documented. It increases skin graft take ratio and speeds up healing. Aim of this study is to compare NPWT to traditional treatment after STSG for any indication in patients aged 18 to 99. This is a two-arm, multicenter, randomized prospective trial with 160 patients.

ELIGIBILITY:
Inclusion Criteria:

* Wound requiring skin graft surgery
* Voluntary

Exclusion Criteria:

* Not voluntary
* Size of wound exceeding 15x15cm or 5x20cm
* Previous skin graft operation to the same wound
* Inability to co-operate
* Wound depth over 1.5cm
* Multiple wounds requiring skin grafting
* Active infection in wound
* Active osteomyelitis in region of wound
* Flap reconstruction of the wound
* Region of wound not suitable for negative pressure wound therapy (for example toes, foot sole)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-09-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Between group difference in skin graft take | 2 weeks after surgery
  Split-thickness skin graft take ratio (percentage of surface area)

SECONDARY OUTCOMES:
Between group difference in skin graft take | 5 to 7 days after surgery
  Split-thickness skin graft take ratio (percentage of surface area)
Between group difference in skin graft take | 8 weeks after surgery
  Split-thickness skin graft take ratio (percentage of surface area)
Strength of pain (wound) | 5 to 7 days after surgery
  Strength of pain in wound (Numeric rating scale 0 to 10; 0= no pain)
Strength of pain (wound) | 2 weeks
  Strength of pain in wound (Numeric rating scale 0 to 10; 0= no pain)
Strength of pain (wound) | 8 weeks after surgery
  Strength of pain in wound (Numeric rating scale 0 to 10; 0= no pain)
Strength of pain (wound) | 1 year after surgery
  Strength of pain in wound (Numeric rating scale 0 to 10; 0= no pain)
Strength of pain (donor site) | 1 week after surgery
  Strength of pain in skin graft donor site (Numeric rating scale 0 to 10; 0= no pain)
Strength of pain (donor site) | 2 weeks after surgery
  Strength of pain in skin graft donor site (Numeric rating scale 0 to 10; 0= no pain)
Strength of pain (donor site) | 8 weeks after surgery
  Strength of pain in skin graft donor site (Numeric rating scale 0 to 10; 0= no pain)
Strength of pain (donor site) | 1 year after surgery
  Strength of pain in skin graft donor site (Numeric rating scale 0 to 10; 0= no pain)
POSAS score (wound) | 8 weeks after surgery
  Patient and Observer Scar Assessment Scale (range 7 to 70 points; 7=best) (wound)
POSAS score (wound) | 1 year after surgery
  Patient and Observer Scar Assessment Scale (range 7 to 70 points; 7=best)(wound)
POSAS score (donor site) | 8 weeks after surgery
  Patient and Observer Scar Assessment Scale (range 7 to 70 points; 7=best) (skin graft donor site)
POSAS score (donor site) | 1 year after surgery
  Patient and Observer Scar Assessment Scale (range 7 to 70 points; 7=best) (skin graft donor site)
Change in quality of life | 5 to7 days after surgery
  Change in EuroQol Group 5-dimension self-report questionnaire (EQ-5D-5L) compared to baseline (before surgery)
Change in quality of life | 2 weeks after surgery
  Change in EuroQol Group 5-dimension self-report questionnaire (EQ-5D-5L) compared to baseline (before surgery)
Change in quality of life | 8 weeks after surgery
  Change in EuroQol Group 5-dimension self-report questionnaire (EQ-5D-5L) compared to baseline (before surgery)
Change in quality of life | 1 year after surgery
  Change in EuroQol Group 5-dimension self-report questionnaire (EQ-5D-5L) compared to baseline (before surgery)
Overall satisfaction | 5 to 7 days after surgery
  Overall satisfaction with treatment (Likert)
Overall satisfaction | 2 weeks after surgery
  Overall satisfaction with treatment (Likert)
Overall satisfaction | 8 weeks after surgery
  Overall satisfaction with treatment (Likert)
Overall satisfaction | 1 year after surgery
  Overall satisfaction with treatment (Likert)
Strength of itching (wound) | 5 to 7 days after surgery
  Strength of itching in wound (Numeric rating scale 0 to 10, 0= no itching)
Strength of itching (wound) | 2 weeks after surgery
  Strength of itching in wound (Numeric rating scale 0 to 10, 0= no itching)
Strength of itching (wound) | 8 weeks after surgery
  Strength of itching in wound (Numeric rating scale 0 to 10, 0= no itching)
Strength of itching (wound) | 1 year after surgery
  Strength of itching in wound (Numeric rating scale 0 to 10, 0= no itching)
Strength of itching (donor site) | 5 to 7 days after surgery
  Strength of itching in skin graft donor site (Numeric rating scale 0 to 10, 0= no itching)
Strength of itching (donor site) | 2 weeks after surgery
  Strength of itching in skin graft donor site (Numeric rating scale 0 to 10, 0= no itching)
Strength of itching (donor site) | 8 weeks after surgery
  Strength of itching in skin graft donor site (Numeric rating scale 0 to 10, 0= no itching)
Strength of itching (donor site) | 1 year after surgery
  Strength of itching in skin graft donor site (Numeric rating scale 0 to 10, 0= no itching)
Length of stay | Until 8 weeks after surgery
  Length of hospital ward stay due to wound treatment (days)
Number of visits | Until 8 weeks after surgery
  Number of visits to hospital due to wound treatment

OTHER OUTCOMES:
Contamination | Immediately before skin graft procedure and antimicrobial prophylaxis
  Type of bacterial flora in wound
Contamination | After revision during skin graft procedure
  Type of bacterial flora in wound
Contamination | 5 to 7 days after skin graft procedure
  Type of bacterial flora in wound

CONTACTS AND LOCATIONS:
Overall Officials: Juha Paloneva, professor, Principal Investigator — Chief medical director
Locations (2):
- Finland (2):
  - Central Finland Hospital, Jyväskylä
  - Tampere University Hospital, Tampere

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serra R, Rizzuto A, Rossi A, Perri P, Barbetta A, Abdalla K, Caroleo S, Longo C, Amantea B, Sammarco G, de Franciscis S. Skin grafting for the treatment of chronic leg ulcers - a systematic review in evidence-based medicine. Int Wound J. 2017 Feb;14(1):149-157. doi: 10.1111/iwj.12575. Epub 2016 Mar 4. PMID 26940940
- [Background] Waltzman JT, Bell DE. Vacuum-assisted closure device as a split-thickness skin graft bolster in the burn population. J Burn Care Res. 2014 Sep-Oct;35(5):e338-42. doi: 10.1097/BCR.0000000000000009. PMID 24577227
- [Background] Blume PA, Key JJ, Thakor P, Thakor S, Sumpio B. Retrospective evaluation of clinical outcomes in subjects with split-thickness skin graft: comparing V.A.C.(R) therapy and conventional therapy in foot and ankle reconstructive surgeries. Int Wound J. 2010 Dec;7(6):480-7. doi: 10.1111/j.1742-481X.2010.00728.x. Epub 2010 Sep 6. PMID 20825510